CLINICAL TRIAL: NCT01090635
Title: Imaging the Uterine Cervix - UltraSightHD™
Status: Completed | Type: Observational
Sponsor: STI-Medical Systems (Industry)
Responsible Party: Rolf Wolters, Sr. VP., STI- Medical Systems
Other Study IDs: 2010-1
Record Dates: First submitted 2010-03-18; First posted 2010-03-22 (Estimated); Last update posted 2011-02-04 (Estimated); Status verified 2011-02

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the performance ability of the UltraSightHD™. The instrument will be assessed on characteristics such as focus quality, ability to image the entire cervix, and illumination. The information gathered from this study will provide data that will be used to determine which settings provide the best imaging outcome for the cervix for a simple screening instrument. Further, this information will serve as the foundation in the development of more advanced follow-on imaging devices.

The primary objectives of this study are to:

* Determine if the light source provides sufficient illumination of the cervix.
* Assess focus and overall image quality.
* Assess the functionality and ergonomics of the instrument's design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Female
* 18 years old or older
* Not pregnant
* Ability to give consent

Exclusion Criteria:

* Male
* Less than 18 years old
* Pregnant or suspected pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy non-pregnant females over 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2010-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Fujita, M.D., Principal Investigator
Locations (1):
- Dr. Nathan Fujita, Honolulu, Hawaii, United States